CLINICAL TRIAL: NCT05900648
Title: Regorafenib and XmAb20717 in Treatment of High-risk Patients With Colorectal Cancer With Radiographic Occult Molecular Residual Disease After End of Established Definitive Therapy (RX-CROME)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 0 participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Xencor, Inc. (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0726; NCI-2023-04464 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Colon Cancer; Rectum Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regorafenib and XmAb20717 (Experimental): Participants will receive regorafenib and XmAb20717 for up to 6 cycles (6 months). Participants will take regorafenib by mouth on Days 1-21 of each cycle. Participants will rest (not take regorafenib) on Days 21-28 of each cycle. Participants will also receive XmAb20717 by vein on Days 1 and 15 of each cycle. Each infusion should take about 60 minutes.
  Interventions: Drug: Regorafenib; Drug: XmAb20717

INTERVENTIONS:
Drug: Regorafenib — Given by PO
  Other Names: BAY 73-4506
Drug: XmAb20717 — Given by (IV) vein

SUMMARY:
To measure the level of circulating tumor DNA (ctDNA) in the blood of colorectal cancer patients after 6 months of receiving therapy with regorafenib and XmAb20717 (also known as vudalimab). ctDNA is genetic material from tumor cells that can be found and measured in the blood

DETAILED DESCRIPTION:
Primary Objective:

1. To determine the 6-month circulating tumor (ctDNA) clearance rate following 6 months of therapy with regorafenib and XmAb20717 (RX regimen) in patients with colorectal cancer (CRC) who present with radiographic occult molecular residual disease (MRD) after completing definitive standard-of-care (SOC) therapy.

Secondary Objectives:

1. To determine the 3-month ctDNA clearance rate following RX treatment.
2. To determine disease-free survival (DFS) following 6 months of RX treatment.
3. To determine overall survival (OS) following 6 months of RX treatment.
4. To determine the safety and tolerability of RX.

Exploratory Objectives:

1. To determine changes in profiles of circulating lymphocytes and ctDNA (including time to ctDNA negative status, duration of ctDNA negative status, overall ctDNA negative rate, lead time from ctDNA detection to radiographic detection) during and following treatment with RX.
2. To determine baseline characteristics in archival tumor and/or plasma that may predict clinical benefit or lack thereof (including but not limited to immune profiles of tumor-infiltrating lymphocytes, expression of immune markers in tumor cells and microenvironment, and tumor molecular profile).

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of CRC
2. Post-R0 resection of stages II, III, or IV CRC and all planned adjuvant therapies have been completed
3. No evidence of radiographic disease within 28 days (before or after) of a positive ctDNA assay
4. Evident MRD as defined by positive ctDNA assay. Patients may be identified for enrollment with any Clinical Laboratory Improvement Amendments (CLIA)-certified ctDNA assay for MRD. MRD status will be confirmed with the Signatera assay prior to initiation of therapy (unless the prior testing was also done with Signatera in which case this test would not require confirmation)
5. Adequate organ and marrow function as defined below:

   1. Absolute neutrophil count: ≥1,000/mcL
   2. Platelets: ≥100,000/mcL
   3. Total bilirubin ≤1.5 x the upper limit of normal (ULN). Total bilirubin (≤3 x ULN) is allowed if Gilbert's syndrome is documented.
   4. AST(SGOT)/ALT(SGPT): ≤3 × institutional ULN (≤5 x ULN for patients with liver involvement of their cancer).
   5. Creatinine clearance ≥40 mL/min. Creatinine clearance (Clcr) can either be measured in a 24-hour urine collection or estimated by the Cockcroft-Gault equation as follows: Clcr (mL/min) = [(140 - age) x (weight in kg) ÷ [72 x (serum creatinine in mg/dL)] [0.85 if female]
6. ECOG performance status (PS) of 0 or 1 (Appendix A)
7. Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of regorafenib in these patients, children <18 years of age are excluded from this study.
8. Able to understand and is willing to sign a written informed consent document.
9. The effects of Regorafenib and XmAb20717 on the developing human fetus are unknown. For this reason and because regorafenib appears to be teratogenic in animal models, women of child-bearing potential (refer to MDA Policy CLN 1114) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for at least 4 months after the last dose. This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure.) Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of administration.

Exclusion Criteria:

1. Concurrent treatment with drug with which the interactions are considered clinically significant by investigator (as outlined in section 5.2). Major surgical procedure or significant traumatic injury within 21 days before start of study medication. Note: If participants received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
2. Systemic therapy with immunosuppressive agents within 7 days or use of any investigational drug within 28 days before the start of trial treatment.
3. Prior exposure to any immune checkpoint blockade agent or any other immunomodulatory agent used for antineoplastic therapy for mCRC.
4. Previous malignant disease (other than the target malignancy to be investigated in this trial) within 3 years prior to study treatment initiation.
5. Receipt of any organ transplantation, including allogeneic stem cell transplantation (exception: transplants that do not require immunosuppression, such as hair transplant).
6. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent.
7. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI-CTCAE v4.03), any history of anaphylaxis, or recent (within 5 months) history of uncontrolled asthma.
8. Clinically significant cardiovascular/ cerebrovascular disease as follows: cerebral vascular accident / stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class >II), or serious cardiac arrhythmia.
9. Clinically relevant diseases (for example, inflammatory bowel disease) and / or uncontrolled medical conditions, which, in the opinion of the Investigator, might impair the subject's tolerance or ability to participate in the trial.
10. Failure to recover from any other toxicity (other than immune-related toxicity) related to previous anticancer treatment to ≤ Grade 2.
11. Receipt of a live-virus vaccine within 30 days prior to first dose of study drug (seasonal flu vaccines that do not contain live virus are permitted).
12. Evidence of any serious bacterial viral (active HIV, HCV or HBV), parasitic, or systemic fungal infections within the 30 days prior to the first dose of study drug.
13. Subject is pregnant or breast feeding or planning to become pregnant while enrolled in the study, up to the final EOT visit.
14. History of (non-infectious) pneumonitis that required steroids, ongoing pneumonitis, or history of interstitial lung disease.
15. Grade > 3 proteinuria ( > 3.5 g/24 hours)
16. Grade > 3 hypertension (systolic blood pressure > 160 or diastolic blood pressure > 100).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kanwal Raghav, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org